CLINICAL TRIAL: NCT06276972
Title: The Relationship Between Spine Coronal Alignment and Lower Limb Biomechanical Parameters in Scoliotic Adolescents. A Cross Sectional Study
Brief Title: Relationship Between Spine Coronal Alignment and Lower Limb Biomechanical in Scoliosis
Status: Active, not recruiting | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ali Elabd, Lecturer of Orthopedic Physical Tehrapy, Delta University for Science and Technology
Other Study IDs: P.T.REC/012/005000
Record Dates: First submitted 2024-02-11; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Scoliosis
Keywords: scoliosis; spine alignment; lower limb; biomechanics
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scoliosis: scoliotic adolescents ranged in age from 10- 18 years will be enrolled
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there's no intervention. it's a cross sectional study correlation study

SUMMARY:
To examine the relationships between spine coronal alignment and lower limb biomechanical parameters in scoliotic adolescents

DETAILED DESCRIPTION:
BACKGROUND:

Adolescent idiopathic scoliosis is one of the most common orthopaedic diseases affecting the spine during adolescence. Numerous studies deal with the aetiology of the disease, X-ray morphology and classification of curvatures and how the disorder disrupts the spinal biomechanical balance, however the disorder is a complex three-dimensional deformity that affects the body as a whole, and these effects must not be overlooked. No cross-section studies were found assessing the connection between sagittal or coronal balance and the biomechanical parameters of the lower extremity.

HYPOTHESES:

Null hypothesis There are no statistically significant relationships between spine coronal alignment and lower limb biomechanical parameters in scoliotic adolescents.

RESEARCH QUESTION:

What are the relationships between spine coronal alignment and lower limb biomechanical parameters in scoliotic adolescents?

PURPOSE: To examine the relationships between spine coronal alignment and lower limb biomechanical parameters in scoliotic adolescents

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with age 10-18 years
* complaining of dorsolumbar scoliosis
* curves (apex lies between D10 and L4)
* curve magnitudes greater than 15 degrees and less than 90
* using or not using brace
* all maturity levels (Risser = 0-5)

Exclusion Criteria:

* Other types of scoliosis ; congenital or neuromuscular
* Current physical therapy or medical treatment for scoliosis,
* Contracture or surgery affecting the lumbar spine or lower limbs
* Pathologies such as inflammatory diseases
* congenital anomalies
* Neurological disorders like cerebral palsy or ataxia
* dislocations
* visual or auditory problems

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: adolescents with idiopathic scoliotic curvature of structural origin and in which any secondary causes could be excluded
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Cobb's angle | at the enrollment
  Cobb's angle for dorso-lumbar scoliosis. The angle of the curve apex from D10 to L4 will be assessed by computed radiograph (X-ray computed scanogram)
Coronal balance | at the enrollment
  Coronal balance estimated by the distance between plumb line and central sacral line from Anetroposterior x-ray view assessed by computed radiograph (X-ray computed scanogram )
length of the the tibia and femur | at the enrollment
  The length (in centimeter) of the Tibia and femur will be assessed by computed radiograph (X-ray computed scan-gram)
tibiofemoral angle | at the enrollment
  The tibiofemoral angle (TFA), or knee angle, is defined as the angle between the anatomical axis of femur with the anatomical axis of tibia. It will be assessed (in degrees) by computed radiograph (X-ray computed scan-gram)
knee joint line convergence angle | at the enrollment
  The knee joint-line convergence angle (KJLCA) h is the angle made by a tangential line between the femoral condyles and the tibial plateau. It will be assessed (in degrees) by computed radiograph (X-ray computed scan-gram)
lower limb mechanical axis; and mechanical axis deviation | at the enrollment
  The mechanical axis of the lower limb, also called the Mikulicz line, is drawn by connecting a point in the center of the femoral head to a point in the center of the ankle. The value of the deviation is measured in millimeters and is named mechanical axis deviation (MAD). It will be assessed by computed radiograph (X-ray computed scan-gram).

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university for science and technology, Gamasa, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
personal preference